CLINICAL TRIAL: NCT06875596
Title: The Effectiveness of an Exercise Program on Scapulohumeral Rhythm, Range of Motion, and Shoulder Girdle Stability in Young Female Handball Players
Brief Title: The Effectiveness of an Exercise Program on Scapulohumeral Rhythm, Range of Motion, and Stability in Young Female Handball Players
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Collaborators: Gdansk College of Health (Unknown)
Responsible Party: Principal Investigator, Bartosz Wilczyński, Principal Investigator, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KB/42/2025
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-03

CONDITIONS: Scapular Dyskinesis; Handball Players; Female Athlete
Keywords: Handball; Sports Performance Assessment; Muscle Strength assessment; Scapular; Scapular dyskinesis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are not informed of the study hypothesis, which is to compare the effects of the upper scapular rotation-based exercise intervention with a standardised upper extremity exercise programme. This will ensure that participants perform to the best of their ability without bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Handball female players (Experimental)
  Interventions: Other: Experimental: Exercise Program
- Control: Handball female players (Active Comparator)
  Interventions: Other: Control: Exercise Program

INTERVENTIONS:
Other: Control: Exercise Program — The entire program begins with an assessment of scapulohumeral rhythm using a digital inclinometer, isometric strength testing, range of motion measurements, the Y-Balance Upper Quarter Test, and the Closed Kinetic Chain Upper Extremity Stability Test. The exercise program for the experimental group lasts eight weeks and is divided into four two-week phases with four sets of exercises targeting the dominant upper extremity only. After the initial assessment, participants will undergo scapular positioning correction for the dominant extremity. They are then introduced to the first set of exercises for the first two weeks. The handball players will be given an exercise sheet explaining each exercise, which they will complete daily after completing their assigned ten minutes of exercise. They will also be given two resistance bands to provide resistance during the assigned exercises. One band is for upper scapular rotation, while the other is for resisting
  Other Names: Control: Handball female players
  Arms: Control: Handball female players
Other: Experimental: Exercise Program — Participants in the active control group will begin the program in the same manner as the experimental group, beginning with scapulohumeral rhythm assessments using a digital inclinometer, isometric strength testing, range of motion measurements, the Y-Balance Upper Quarter Test, and the Closed Kinetic Chain Upper Extremity Stability Test. They will also follow an eight-week exercise program divided into four two-week phases with four sets of exercises targeting the dominant upper extremity only. The key difference is that the control group will not focus on correcting scapular position for upward rotation during the exercises. Specifically, they will skip the upward rotation exercises at the beginning of each set and will not incorporate the acquired upward rotation control into other movement exercises. You will also be given a resistance band to provide resistance during the assigned exercises.
  Other Names: Experimental: Handball female players Exercise Program
  Arms: Experimental: Handball female players

SUMMARY:
The primary objective of this study is to investigate the effectiveness of a shoulder girdle exercise program in improving stability, range of motion, and motor control in female handball players.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of a structured shoulder girdle exercise programme on stability, range of motion (ROM) and motor control in female handball players. The study will be conducted over a period of 8 weeks and will involve 60 participants aged 17-30 years recruited from professional handball clubs. Participants will be randomly assigned to either the experimental group, which will follow a modified version of the Watson programme, or the control group, which will continue with their standard training programme. Aims: - To compare the effects of the upper scapular rotation-oriented exercise intervention with a standardised upper extremity exercise programme. - Scapulohumeral rhythm assessment: To assess scapulohumeral rhythm at different angles of shoulder flexion (30°, 60°, 90° and 120°) in young female handball players, with a focus on identifying potential asymmetries between the dominant and non-dominant limbs. - Analysis of scapular kinematics: To measure scapular upward rotation, anterior/posterior tilt and medial/lateral translation at different degrees of shoulder flexion to identify movement patterns associated with scapular dyskinesis. - Functional stability analysis: To assess upper extremity functional stability using the Y-Balance Upper Quarter Test (YBT-UQ) and the Closed Kinetic Chain Upper Extremity Stability Test pre- and post-exercise to identify potential correlations between stability improvements and changes in scapular rhythm and muscle activation. - Isometric strength measurement: To evaluate isometric strength in shoulder abduction, internal rotation and external rotation using the Lafayette HHD handheld dynamometer to assess the impact of the intervention on shoulder muscle performance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals with no reported health problems
* No history of shoulder or elbow surgery within the past 2 years
* Received information about the study
* Written consent from the participant to participate in the study, including video recording and photography

Exclusion criteria:

* Injury or trauma to the upper extremity within the past 3 months
* Illness that prevents participation in the study or tests
* Heavy physical activity of the shoulder girdle within 2 hours prior to the study
* Orthopedic surgery or physiotherapy treatment of the shoulder girdle

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-08 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2028-02-10 (Estimated)

PRIMARY OUTCOMES:
Scapulohumeral rhythm | through study completion, an average of 2 years
  Scapular upward rotation is assessed with the Digital Inclinometer (BASELINE 12-1057) in a seated position to minimize compensatory movements of the trunk and lower extremities. The first measurement is taken at baseline (0° of shoulder flexion), followed by additional measurements at 30°, 60°, 90°, and 120° of shoulder flexion. Each position is held for 10-15 seconds to ensure stable measurement conditions. Measurements are repeated three times and the average is used for analysis. The assessment will be performed on both the dominant and non-dominant upper limb to evaluate movement symmetry. Data will be recorded manually by a research assistant to reduce the risk of reading errors and to ensure measurement accuracy. Statistical analysis will be performed to determine the scapulohumeral rhythm across different ranges of motion and to identify potential movement asymmetries.
ISOMETRIC STRENGTH TEST - Internal and External Rotation | through study completion, an average of 2 years
  Isometric strength assessment of the shoulder girdle muscles will be conducted using the Lafayette Hand-Held Dynamometer (HHD). For the rotator muscles, measurements will be performed in the prone position with the shoulder abducted to 90° and the elbow flexed to 90°, with the forearm hanging freely over the edge of the examination table. This setup will be used for both internal and external rotation strength assessments. Results are expressed in Newtons (N) or normalized to body weight as Newtons per kilogram (N/kg).
Y-Balance Upper Quarter Test (YBT-UQ) | through study completion, an average of 2 years
  The Y-Balance Upper Quarter Test (YBT-UQ) is used to assess upper extremity stability and reach performance. The test requires the participant to maintain a single-arm support position while the opposite arm performs reaching movements in three directions: anterior (forward), inferolateral (diagonally opposite the supporting hand), and superolateral (diagonally toward the supporting hand).
  Each reach is measured in centimeters, and the final score for each direction is calculated as the average of three trials. The test will be performed on both upper limbs and arm length will be included in the analysis to ensure standardized results. Results will be reported in centimeters, "cm", and Upper Limb Length % (standardized by upper limb length).

SECONDARY OUTCOMES:
RANGE OF MOTION (Shoulder Internal and External Rotation) | through study completion, an average of 2 years
  Range of motion is measured for internal and external rotation of the shoulder. The participant is positioned in the prone position with the shoulder abducted to 90 degrees and the elbow flexed to 90 degrees, allowing the forearm to hang freely over the edge of the examination table. The starting position (0 degrees) is defined as the forearm being vertically aligned. Results are presented in degre
Closed Kinetic Chain Upper Extremity Stability Test | through study completion, an average of 2 years
  Two strips of tape will be placed on the floor 90 cm apart. Participants will be instructed to assume a push-up position and perform as many hand touches as possible on each strip within 15 seconds. The examiner will count the number of touches.
  Three trials will be conducted, and the final score will be calculated as the average number of touches across all three trials. A 45-second rest period will be provided between each trial.
  The CKCUEST score and CKCUEST power will be calculated using the following formulas:
  * Score = Average number of touches on CKCUEST / height (m)
  * Power = 68% of body weight (kg) × Average number of touches on CKCUEST

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Immunobiology and Environment Microbiology, Medical University of Gdańsk, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided